CLINICAL TRIAL: NCT05153590
Title: Weight Loss and Treatment Patterns in a Real World Population of Adults Receiving Saxenda® for Weight Management in Routine Clinical Practice in Switzerland
Brief Title: A Research Study About Weight Loss and Treatment Patterns With the Use of Saxenda® in Adults in Real-life Settings in Switzerland
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8022-4823; U1111-1263-5715 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-11-30; First posted 2021-12-10 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-09

CONDITIONS: Obesity or Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reimbursed: The reimbursed cohort includes only patients who received Saxenda® through mandatory basic insurance
  Interventions: Drug: Saxenda®
- Non reimbursed: The non reimbursed cohort includes patients who received Saxenda® through additional private insurance or self-pay
  Interventions: Drug: Saxenda®

INTERVENTIONS:
Drug: Saxenda® — Patients will be treated with commercially available Saxenda® according to local label and to routine clinical practice at the discretion of the treating physician.
  The indication is for adults who need help managing their weight based on two different body mass index (BMI) groups.

SUMMARY:
The study is investigating weight loss and treatment patterns associated with the use of Saxenda® in adult patients.

The aim of the study is to assess the weight loss associated with Saxenda® in patients with obesity or overweight. Saxenda® was prescribed to participants by study doctor independently of this study.

The study will last for about 4 months, where the data will be collected from the available medical records.

There will be no additional activities expected from participants in the scope of study because it is a chart-review study.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent (general consent for research or study-specific informed consent) obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female, aged 18 to 74 years (both inclusive) at the time of Saxenda® initiation.
* Have been prescribed Saxenda® for weight management.
* For the reimbursed cohort, per the Swiss reimbursement criteria: BMI greater than or equal to 35 kg/m^2 or a BMIgreater than or equal to 28 and below 35 kg/m^2 with additional weight related comorbidities (pre diabetes or T2D (Type 2 Diabetes Mellitus), hypertension, dyslipidaemia), prior to receiving the Saxenda® treatment.
* For the non-reimbursed cohort, BMI greater than or equal to 30 kg/m^2 or a BMI greater than or equal to 28 kg/m^2 with additional weight related comorbidities (pre diabetes or T2D, arterial hypertension, dyslipidaemia), prior to receiving the Saxenda® treatment.
* The decision to initiate treatment with commercially available Saxenda® has been made by the patient/legally acceptable representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.
* Baseline weight measurement within 3 months of Saxenda® initiation/prescription.
* At least one weight assessment post-Saxenda® initiation/prescription.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Treatment with any investigational drug within 30 days of Saxenda® prescription/initiation.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Concomitant treatment of Saxenda® with other GLP 1 (Glucagon-like peptide-1) receptor agonists, or orlistat.
* Concomitant treatment with sodium/glucose cotransporter-2 inhibitors (SGLT 2i), dipeptidyl peptidase-4 (DPP 4i), or insulin for the reimbursed cohort only.
* Patients who have been treated with any obesity medication for last 12 weeks prior to initiation of Saxenda® treatment.
* Patients who have previously been treated with a GLP 1 receptor agonist for the reimbursed cohort only.
* Patients who have undergone bariatric surgery at any time before starting Saxenda® treatment.
* Patients initiating Saxenda® treatment after 31 October 2020.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of male or female adults who have been prescribed Saxenda® for weight management in 2 cohorts reimbursed and non reimbursed
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Relative change in body weight greater than or equal to 5% (lower BMI with weight related comorbidities) or greater than or equal to 7% (higher BMI) in reimbursed setting (yes/no) | From Baseline (Week 0) to Week 16
  Percentage of patients - yes
Relative change in body weight greater than or equal to 5%, conditionally to relative change greater than or equal to 5% or greater than or equal to 7% at Week 16 in reimbursed setting(yes/no) | From Week 16 to Month 10
  Percentage of patients - yes

SECONDARY OUTCOMES:
Reimbursed setting: Absolute change in body weight | From Baseline (Week 0) to Week 16
  messured in kg
Reimbursed setting: Relative change in body weight | From Baseline (Week 0) to Week 16
  messured in percent
Reimbursed setting: Absolute change in body weight | From Week 16 to Month 10
  messured in kg
Reimbursed setting: Relative change in body weight | From Week 16 to Month 10
  messured in percent
Reimbursed setting: Absolute change in body weight | From Baseline (Week 0) to Month 10
  messured in kg
Reimbursed setting: Relative change in body weight | From Baseline (Week 0) to Month 10
  messured in percent
Reimbursed setting: Time on Saxenda® | From Baseline (Week 0) to end of study date
  messured in day
Reimbursed setting: Discontinuation of patient (yes/no) | From Baseline (Week 0) to Week 16
  Percentage of patients - yes/no
Reimbursed setting: Discontinuation of patient (yes/no) | From Week 16 to Month 10
  Percentage of patients - yes
Reimbursed setting: Discontinuation of patient (yes/no) | From Baseline (Week 0) to Month 10
  Percentage of patients - yes
Reimbursed setting: Presence of obesity-related comorbidities identified by authorities (*pre-diabetes, type 2 diabetes, dyslipidaemia and hypertension) | Baseline
  Percentage of patients - yes
Non-reimbursed setting: Time on Saxenda® | From Baseline (Week 0) to end of study date
  messured in Day
Non-reimbursed setting: Discontinuation of patient (yes/no) | From Baseline (Week 0) to Week 16
  Percentage of patients - yes
Non-reimbursed setting: Discontinuation of patient (yes/no) | From Week 16 to Month 10
  Percentage of patients - yes
Non-reimbursed setting:Discontinuation of patient (yes/no) | From Baseline (Week 0) to Month 10
  Percentage of patients - yes
Non-reimbursed setting: Discontinuation of patient (yes/no) | From Baseline (Week 0) to end of study date
  Percentage of patients - yes
Non-reimbursed setting: Presence of obesity-related comorbidities identified by the authorities (pre-diabetes, type 2 diabetes, dyslipidaemia and hypertension) | Baseline
  Percentage of patients - yes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Soeborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com